CLINICAL TRIAL: NCT03620318
Title: Compassionate Use of Crenolanib for Cancers With Platelet Derived Growth Factor Receptor Alpha (PDGFRa) Mutations, PDGFRa Amplifications or Fms-like Tyrosine Kinase 3 (FLT3) Mutations
Brief Title: Individual Patient Compassionate Use of Crenolanib
Status: Available | Type: Expanded Access
Sponsor: Arog Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ARO-EAP
Record Dates: First submitted 2018-08-02; First posted 2018-08-08 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: FLT3-ITD Mutation; FLT3/TKD Mutation; PDGFR-Alpha D842V; PDGFRA Gene Amplification
Keywords: Compassionate use

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Crenolanib besylate

SUMMARY:
Compassionate use of crenolanib for patients with serious life-threatening illness that have exhausted all available therapies used to treat the disease, with no other viable therapy options, who is not eligible for clinical trials. This program is designed to evaluate the requests on a patient by patient basis.

Patients must have documented evidence of a point mutation in position 842 in platelet derived growth factor receptor alpha (PDGFRA-D842V) or amplification of PDGFRA or internal tandem duplication within the FMS-like tyrosine kinase 3 (FLT3-ITD) or point mutations within the tyrosine kinase domain (TKD) of FLT3 (FLT3-TKD)

DETAILED DESCRIPTION:
This program is being offered on a patient by patient basis while phase 3 studies with crenolanib are ongoing.

Institutional Review Board-/Independent Ethics Committee approval must be granted before, The experimental intervention will be administered over 28-day cycles. Compassionate use of crenolanib will be limited such that it does not interfere with the supply need for phase 3 studies.

There must be adequate understanding of the indication for the requested use.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have a serious life threatening cancer with FLT3/PDGFRa mutation or PDGFRa amplification who has exhausted all other treatment options
* Subject and their partner (if adults) must use 2 forms of contraception during study and for 3 months following last dose of study drug

Exclusion Criteria:

* Subject is eligible for enrollment in an ongoing clinical trial
* Subject has any condition which, in the investigator's opinion makes the subject unsuitable for participation

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Policlinico San Martino, Genova, Italy